CLINICAL TRIAL: NCT06558942
Title: A Study on the Application of Incisional Negative Pressure Therapy in Reducing the Risk of Infection in Animal Induced Injury Patients With Primary Wound Closure
Brief Title: Incisional Negative Pressure Therapy to Prevent Animal Induced Wound Infection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024SF59
Record Dates: First submitted 2024-08-11; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Injury Caused by Animal Bites; Wound Infection
Keywords: Animal bite injury; Incision negative pressure treatment technology; Wound infection rate
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- iNPWT group (Experimental): The clinical data of 60 patients who met the inclusion and exclusion criteria were collected prospectively, including: gender, age, smoking, body mass index (BMI), hypertension, diabetes, aspirin and other antiplatelet drugs, anticoagulants, injured animals (dogs or cats), wound parameters (including wound site, wound length, wound depth, and time of subsequent diagnosis). Rinse the patient's wound with a weak alkaline disinfectant for 15 minutes, thoroughly clean the wound, and then suture it in one stage. Place the device of incisional negative pressure wound therapy (iNPWT) and evaluate the wound quality for 2-3 days. If necessary, extend the use of the iNPWT device. All patients received prophylactic use of antibiotics within one week.
  Interventions: Device: incisional negative pressure wound technology

INTERVENTIONS:
Device: incisional negative pressure wound technology — Negative pressure device used directly on closed or sutured incisions
  Other Names: iNPWT

SUMMARY:
Animal injuries are a significant public health issue, with the most common being bites or scratches from cats and dogs. Every year, over 40 million people in China are bitten or scratched by cats and dogs, which can lead to wound infections and even systemic complications, with infection rates ranging from 10% to 80%. However, there is still no better way to reduce wound infection rates in current clinical studies and guidelines.

Incisional negative pressure wound therapy (iNPWT) is a new wound treatment technology developed in recent years. It creates a negative pressure environment on sutured or closed wounds, helps to fix the edges of the incision together, reduce lateral tension on the wound, stimulate blood perfusion at the edge of the wound, remove fluid from the wound, and act as an external pollution barrier. INPWT has been widely used for postoperative wound healing in surgery, but there is currently a lack of effective clinical trials on its ability to prevent wound infections caused by animal injuries and promote wound healing.

This study aims to apply iNPWT technology to the wounds of patients with rabies grade III exposure who underwent primary suturing, and compare it with wounds covered with ordinary gauze after previous primary suturing to determine whether it can help reduce postoperative incision infection rates and promote wound healing. This will provide high-quality clinical evidence for the widespread use of wound management in rabies grade III exposure patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Limds injuries caused by animals, first or second animal injury to Grade III exposed patients, with deep wounds reaching the fat layer, tendons, and even penetrating injuries.
* Patients with wounds>2cm and severe injuries that even require surgical treatment.

Exclusion Criteria:

* Missing or incomplete follow-up data within 30 days.
* Patients who have been infected with wounds or have been injured for more than 8 hours before seeking medical attention.
* Acupuncture like wound (<2mm).
* Patients with whole skin detachment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Wound infection (WI) | <4 weeks
  The local skin of the wound appears red, swollen, hot, and painful, with or without systemic hyperthermia

SECONDARY OUTCOMES:
Delayed healing of wounds (DHW) | 2-4 weeks
  Wound healing time is longer than 14 days.
Wound reprocessing (WR) | ≤4 weeks
  Including wound dehiscence, hematoma, seroma and other situation needed to switch treatments.
other wound complication | ≤4 weeks
  redness and rash of skin around the wound.

CONTACTS AND LOCATIONS:
Overall Officials: Shi Jiping, Master, Principal Investigator — Peking University First Hospital
Locations (1):
- Emergency Department of Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen F, Liu Q, Jiang Q, Shi J, Luba TR, Hundera AD, Fang P, Cao S, Lu Z. Risk of human exposure to animal bites in China: a clinic-based cross-sectional study. Ann N Y Acad Sci. 2019 Sep;1452(1):78-87. doi: 10.1111/nyas.14202. Epub 2019 Aug 9. PMID 31397929
- [Result] Philipsen TE, Molderez C, Gys T. Cat and dog bites. What to do? Guidelines for the treatment of cat and dog bites in humans. Acta Chir Belg. 2006 Nov-Dec;106(6):692-5. doi: 10.1080/00015458.2006.11679983. PMID 17290697
- [Result] Fernandez Vecilla D, Aspichueta Vivanco C, Ugalde Zarraga E, Diaz de Tuesta Del Arco JL. Wound infection caused by Pasteurella canis and Neisseria animaloris after a dog bite. Rev Esp Quimioter. 2023 Dec;36(6):635-637. doi: 10.37201/req/035.2023. Epub 2023 Sep 29. No abstract available. PMID 37772341
- [Result] Eichenauer F, Kim S, Hakimi M, Eisenschenk A, Weber S. [Infections of the Hand after Bite Injuries]. Handchir Mikrochir Plast Chir. 2021 Jun;53(3):237-244. doi: 10.1055/a-1382-8093. Epub 2021 Jun 16. German. PMID 34134156
- [Result] Zangari A, Cerigioni E, Nino F, Guidi R, Gulia C, Piergentili R, Ilari M, Mazzoni N, Cobellis G. Dog bite injuries in a tertiary care children's hospital: A seven-year review. Pediatr Int. 2021 May;63(5):575-580. doi: 10.1111/ped.14484. Epub 2021 Apr 20. PMID 32979010
- [Result] Miller C. The History of Negative Pressure Wound Therapy (NPWT): From "Lip Service" to the Modern Vacuum System. J Am Coll Clin Wound Spec. 2013 Nov 28;4(3):61-2. doi: 10.1016/j.jccw.2013.11.002. eCollection 2012 Sep. PMID 26236637
- [Result] Fleischmann W, Strecker W, Bombelli M, Kinzl L. [Vacuum sealing as treatment of soft tissue damage in open fractures]. Unfallchirurg. 1993 Sep;96(9):488-92. German. PMID 8235687
- [Result] Morykwas MJ, David LR, Schneider AM, Whang C, Jennings DA, Canty C, Parker D, White WL, Argenta LC. Use of subatmospheric pressure to prevent progression of partial-thickness burns in a swine model. J Burn Care Rehabil. 1999 Jan-Feb;20(1 Pt 1):15-21. doi: 10.1097/00004630-199901001-00003. PMID 9934631
- [Result] Stannard JP, Robinson JT, Anderson ER, McGwin G Jr, Volgas DA, Alonso JE. Negative pressure wound therapy to treat hematomas and surgical incisions following high-energy trauma. J Trauma. 2006 Jun;60(6):1301-6. doi: 10.1097/01.ta.0000195996.73186.2e. PMID 16766975
- [Result] Glaser DA, Farnsworth CL, Varley ES, Nunn TA, Sayad-Shah M, Breisch EA, Yaszay B. Negative pressure therapy for closed spine incisions: a pilot study. Wounds. 2012 Nov;24(11):308-16. PMID 25876166
- [Result] De Leon JC, Karia RA. Incisional and Surrounding Periarticular Soft Tissue Management With Negative Pressure Therapy. J Orthop Trauma. 2022 Sep 1;36(Suppl 4):S26-S30. doi: 10.1097/BOT.0000000000002429. PMID 35994306
- [Result] Dohmen PM, Misfeld M, Borger MA, Mohr FW. Closed incision management with negative pressure wound therapy. Expert Rev Med Devices. 2014 Jul;11(4):395-402. doi: 10.1586/17434440.2014.911081. Epub 2014 Apr 22. PMID 24754343
- [Result] Gabriele L, Gariffo G, Grossi S, Ipponi E, Capanna R, Andrean L. Closed Incisional Negative Pressure Wound Therapy (ciNPWT) in Oncological Orthopedic Surgery: Preliminary Report. Surg Technol Int. 2021 May 20;38:451-454. doi: 10.52198/21.STI.38.OS1429. PMID 33755942
- [Result] Newman JM, Siqueira MBP, Klika AK, Molloy RM, Barsoum WK, Higuera CA. Use of Closed Incisional Negative Pressure Wound Therapy After Revision Total Hip and Knee Arthroplasty in Patients at High Risk for Infection: A Prospective, Randomized Clinical Trial. J Arthroplasty. 2019 Mar;34(3):554-559.e1. doi: 10.1016/j.arth.2018.11.017. Epub 2018 Nov 17. PMID 30545653
- [Result] Salmenkyla T, Kilpivaara K, Ohtonen P, Rautio T, Makarainen E. Case control study investigating the clinical utility of NPWT in the perineal region following abdominoperineal resection for rectal adenocarcinoma: a single center study. BMC Surg. 2022 Jul 30;22(1):296. doi: 10.1186/s12893-022-01746-1. PMID 35907824
- [Result] Mehdorn M, Niebisch S, Scheuermann U, Gockel I, Jansen-Winkeln B. Incisional negative pressure wound therapy does not reduce surgical site infections in abdominal midline incisions: a case control study. Acta Chir Belg. 2020 Aug;120(4):250-256. doi: 10.1080/00015458.2019.1599180. Epub 2019 Apr 12. PMID 30975040
- [Result] Groenen H, Jalalzadeh H, Buis DR, Dreissen YEM, Goosen JHM, Griekspoor M, Harmsen WJ, IJpma FFA, van der Laan MJ, Schaad RR, Segers P, van der Zwet WC, de Jonge SW, Orsini RG, Eskes AM, Wolfhagen N, Boermeester MA. Incisional negative pressure wound therapy for the prevention of surgical site infection: an up-to-date meta-analysis and trial sequential analysis. EClinicalMedicine. 2023 Jul 24;62:102105. doi: 10.1016/j.eclinm.2023.102105. eCollection 2023 Aug. PMID 37538540